CLINICAL TRIAL: NCT07096947
Title: A Multifactor Prediction Model for Non-curative Outcomes in Mixed-type Early Gastric Cancer: a Retrospective Cohort Study
Brief Title: A Multifactor Prediction Model for Non-curative Outcomes in Mixed-type Early Gastric Cancer
Acronym: MTEGC
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Lu Han, Principal Investigator, The First Affiliated Hospital of Nanchang University
Other Study IDs: FirstNanchangU-97696617; 82360112 (Other Grant/Funding Number: the National Natural Science Foundation of China); 2024A0032 (Other Grant/Funding Number: Jiangxi Provincial Traditional Chinese Medicine Administration Science and Technology Plan)
Record Dates: First submitted 2025-07-08; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Mixed-type Early Gastric Cancer
Keywords: Mixed-type Early Gastric Cancer; Non-curative Outcomes; Nomogram Model; Prognosis; Dual-center Retrospective Cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A training set: The patients with early gastric cancer (EGC) who underwent radical gastrectomy at the Donghu Ward of the First Affiliated Hospital of Nanchang University
- A internal validation set: The patients with early gastric cancer (EGC) who underwent radical gastrectomy at the Xianghu Ward of the First Affiliated Hospital of Nanchang University
- A external validation set: The patients with early gastric cancer (EGC) who underwent radical gastrectomy of the Second Affiliated Hospital of Nanchang University

SUMMARY:
The goal of this dual-center study is to identify the most valuable predictive factors (MVPs) for non-curable mixed-type early gastric cancer (NC-MTEGC) and develop a nomogram scoring model to assist surgeons in formulating precise postoperative combined radiochemotherapy strategies in patients with mixed-type early gastric cancer (MTEGC) who have undergone radical surgical resection. The main question it aims to answer is:

What are the most valuable predictive factors for NC-MTEGC, and can a nomogram scoring model developed based on these factors effectively assist in formulating precise postoperative combined radiochemotherapy strategies?

Patients with MTEGC who have undergone radical surgical resection (including 160 in the training group, 151 in the internal validation set from the First Affiliated Hospital of Nanchang University, and 110 in the external test cohort from the Second Affiliated Hospital of Nanchang University) will be included in the study. The Least Absolute Shrinkage and Selection Operator (LASSO) algorithm will be used to assess key predictive indicators, a nomogram prediction model will be developed based on logistic regression, and an NC-MTEGC risk score model will be constructed. Meanwhile, the model's discriminatory ability, calibration, and clinical utility will be comprehensively validated across the three cohorts, with follow-up for relevant conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Mixed-type early gastric cancer (MTEGC);
2. Receive a surgical procedure;
3. Complete preoperative data.

Exclusion Criteria:

1. Received neoadjuvant therapy;
2. History of gastrectomy;
3. Previous cancer or residual gastric cancer (GC);
4. Distant metastasis at diagnosis;
5. Incomplete preoperative data;
6. Undifferentiated MTEGC components;
7. Missing imaging data or refusal of follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: mixed-type early gastric cancer
Sampling Method: Non-Probability Sample
Enrollment: 421 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse postoperative prognosis in patients with mixed-type early gastric cancer | From enrollment to the end of treatment at 5 years
  Evaluate the incidence of adverse postoperative prognosis in patients with mixed-type early gastric cancer via the Nomogram model scoring.

SECONDARY OUTCOMES:
Pathological malignancy grade | Periprocedural
  Grading criteria refer to clinical guidelines: High risk, Medium risk, Low risk.

OTHER OUTCOMES:
Lymph node metastasis detected by CT | From enrollment to the end of treatment at 5 years
  The status of lymph node metastasis is divided into "no lymph node metastasis (no tumor cell invasion of lymph nodes detected)" and "lymph node metastasis (the presence of tumor cell invasion of lymph nodes)".
Tumor lesion long diameter | Periprocedural
  Measured and reported in millimeters (mm)
Ulcer long diameter | Periprocedural
  Measured and reported in millimeters (mm)
T stage | Periprocedural
  Staging criteria refer to clinical guidelines
Gender | Baseline
  Binary classification, divided into male and female
Ki67 expression level | Periprocedural
  Measured and reported as a percentage (%)
P53 expression level | Periprocedural
  Measured and reported as a percentage (%)
Lesion location | Periprocedural
  The lesion locations are classified as follows: Gastric Body, Gastric Antrum, Gastric Angle, Cardia, Pylorus, and Antrum-Body Junction.
CEA level | Baseline
  Measured and reported in nanograms per milliliter (ng/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No
The secure sharing of Individual Participant Data (IPD) must adhere to the principles of "privacy protection first, minimum necessity, and full-process controllability". It should integrate technical safeguards (such as de-identification and encryption), management norms (including access control and protocol constraints), and compliance reviews. This approach aims to promote collaboration in medical research while maximizing the protection of participants' rights and interests.